CLINICAL TRIAL: NCT04424667
Title: Clinical and Economic Impact of Supplementation With Donor Milk Pasteurized by HTST Method Versus Holder Method in Extremely Birth Weight Preterm Infants. Randomized Clinical Trial
Brief Title: Clinical Impact of Donor Milk Pasteurized by HTST Treatment in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmen Rosa Pallas (Other)
Responsible Party: Sponsor-Investigator, Carmen Rosa Pallas, Head of Neonatology Service, MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Neo-HTST
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Late-Onset Neonatal Sepsis
Keywords: neonatal sepsis; extremely low birth weight infant; donor milk; HTST pasteurization; Holder pasteurization
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holder pasteurization (Active Comparator): Donor milk pasteurized by Holder method (62.5ºC, 30 minutes)
  Interventions: Other: donor milk
- HTST pasteurization (Experimental): Donor milk pasteurized by High Temperature Short Time (HTST) method (72ºC, 15 seconds)
  Interventions: Other: donor milk

INTERVENTIONS:
Other: donor milk — pasteurized donor milk

SUMMARY:
Randomized double-blind clinical trial to compare the incidence of microbiological proven late onset sepsis in extremely preterm infants (<1000 grams) that are supplemented with donor milk pasteurized by High Temperature Short Time (HTST) method versus the Holder method.

DETAILED DESCRIPTION:
Donor milk pasteurized by an innovative High Temperature Short Time (HTST) system (patented by researchers) retains more immune and trophic compounds than pasteurized milk by traditional Holder method. These compounds are related to the protection conferred by breast milk against nosocomial sepsis and necrotizing enterocolitis in preterm infants, so it would be of interest to study if there is a clinical benefit in these patients when health professionals are supplementing with donor milk pasteurized by both methods.

The purpose of this study is to compare the incidence of microbiological proven late onset sepsis in newborns under 1000 grams that in the first 28 days of life need to be supplemented with donor milk pasteurized by HTST method versus the Holder method.

This is a randomized double-blind clinical trial with parallel assignment. A total of 305 premature babies with a birth weight of less than 1000 grams will be recruited, admitted to the Neonatology Services of the Hospital 12 de Octubre and the Hospital de La Paz and meet the inclusion criteria. Half of the patients will be supplemented exclusively with donor milk pasteurized by the HTST system and the other half with pasteurized milk by the Holder method. Linear generalized models will be used for longitudinal data analysis.

ELIGIBILITY:
Inclusion Criteria (all criteria are necessary) :

* Infants weighing 1000 grams or less at birth
* Infants born or transferred before the third day of life to the participating centers
* Start enteral feeding in the first week of life
* Receive any amount of donor milk in the first 28 days of life
* Informed consent signed by parents or legal guardians

Exclusion Criteria:

* Language barrier
* Infants with chromosomopathies
* Infants with major congenital malformations
* Infants with severe asphyxiation (cord pH or first arterial pH <7)
* Infants included in another clinical trial that modifies nutritional management
* Infants who previously fed with formula

Post-randomization exclusion criteria:

- Randomized infant who do not fulfill inclusion criteria

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Microbiological proven late onset sepsis rate | From the time and day of randomization until the date of discharge from the neonatal unit, assessed up to 24 weeks
  Incidence of Microbiological proven late onset sepsis expressed as a percentage

SECONDARY OUTCOMES:
Central line associated bloodstream infections (CLABSI) rate | From the time and day of randomization until the date of discharge from the neonatal unit, assessed up to 24 weeks
  Number of CLABSI events per 1000 catheter-days
Necrotizing enterocolitis (NEC) and/or microbiological proven late onset sepsis rate | From the time and day of randomization until the date of discharge from the neonatal unit, assessed up to 24 weeks
  Incidence of NEC nad late onset sepsis as a percentage
Mortality rate | From the time and day of randomization until the date of discharge from the neonatal unit, assessed up to 24 weeks
  Percentage of preterm infant died during the study
Oxygen supplementation | Assessed up to 24 weeks
  Percentage of infants with respiratory assistance with fraction of inspired oxygen greater than 0.21 at 36 weeks postmenstrual age
Stage 3-5 Retinopathy | From the time and day of randomization until the date of discharge from the neonatal unit, assessed up to 24 weeks
  Percentage of infants diagnosed with retinopathy by the ophthalmologist
Growth velocity | Assessed up to 24 weeks
  Growth calculated as the weight gain in g/kg/day

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Rosa Pallas Alonso, Study Chair — Hospital Universitario 12 de Octubre
Locations (2):
- Spain (2):
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No